CLINICAL TRIAL: NCT01844284
Title: A Clinical Evaluation of AVJ-301 (Absorb™ BVS), the Everolimus Eluting Bioresorbable Vascular Scaffold in the Treatment of Subjects With de Novo Native Coronary Artery Lesions in Japanese Population
Brief Title: AVJ-301 Clinical Trial: A Clinical Evaluation of AVJ-301 (Absorb™ BVS) in Japanese Population
Acronym: ABSORB JAPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-301
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Absorb™ BVS; Angioplasty; Bioabsorbable; Bioreabsorbable; BVS; Coronary Artery Disease; Coronary Artery Endothelial Responsiveness; Coronary artery restenosis; Coronary artery stenosis; Coronary scaffold; Coronary Stent; Drug eluting stents; Everolimus; Myocardial ischemia; Stent thrombosis; Stents
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Restenosis; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorb™ BVS (Experimental): Subjects receiving Absorb™ BVS
  Interventions: Device: Absorb™ BVS
- XIENCE PRIME®/XIENCE Xpedition™ (Active Comparator): Subjects receiving XIENCE PRIME®/XIENCE Xpedition™
  Interventions: Device: XIENCE PRIME®/XIENCE Xpedition™

INTERVENTIONS:
Device: XIENCE PRIME®/XIENCE Xpedition™ — Subjects receiving XIENCE PRIME®/XIENCE Xpedition™
  Arms: XIENCE PRIME®/XIENCE Xpedition™
Device: Absorb™ BVS — Subjects receiving Absorb™ BVS
  Arms: Absorb™ BVS

SUMMARY:
Prospective, Randomized (2:1), active control, single-blind, non-inferiority, multicenter, Japanese Clinical Trial to evaluate the safety and effectiveness of Absorb™ BVS (AVJ-301) in the treatment of subjects with ischemic heart disease caused by de novo native coronary artery lesions in Japanese population by comparing to approved metallic drug eluting stent.

DETAILED DESCRIPTION:
Absorb™ BVS is currently in development at Abbott Vascular. Not available for sale in the US or Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 20 years of age.
2. Subject or a legally authorized representative must provide written Informed Consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia) suitable for elective percutaneous coronary intervention (PCI).
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must be able to take dual antiplatelet therapy for up to 1 year following the index procedure and anticoagulants prior/during the index procedure. Therefore the subject has no known allergic reaction, hypersensitivity or contraindication to aspirin, clopidogrel, ticlopidine or heparin.
6. Female subject of childbearing potential must not be pregnant* at the index procedure and does not plan pregnancy for up to 1 year following the index procedure.

   * Except for non-pregnancy is apparent, negative pregnancy result within 7 days prior to the index procedure is required.
7. Female subject is not breast-feeding at the time of the screening visit and will not be breast-feeding for up to 1 year following the index procedure.
8. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 13 months following the index procedure

Exclusion Criteria:

1. Elective surgery is planned within 1 year after the procedure that will require general anesthesia or discontinuing either aspirin or Thienopyridine.
2. Subject has known hypersensitivity or contraindication to device material and its degredants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated.
3. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
4. Subject had an acute myocardial infarction (AMI) within 72 hours of the index procedure

   * The subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes
   * Creatine Kinase (CK) and Creatine Kinase - Muscle and Brain (CK-MB) have not returned to within normal limits at the time of index procedure.
5. Subject has an unstable cardiac arrhythmia which is likely to become hemodynamically unstable due to arrhythmia.
6. Subject has a known left ventricular ejection fraction (LVEF) < 30% (LVEF may be obtained at the time of the index procedure if the value is unknown and the investigator believes it is necessary).
7. The target vessel was treated by PCI within 12 months.
8. Prior PCI within the non-target vessel is acceptable if performed anytime > 30 days before the index procedure or between 24 hours and 30 days before the index procedure if successful and uncomplicated.
9. Subject requires future staged PCI either in target or non target vessels.
10. Subject has a malignancy that is not in remission.
11. Subject is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.,). Note: corticosteroids are not included as immunosuppressant therapy, diabetes mellitus is not regarded as autoimmune disease.
12. Subject has received any solid organ transplants or is on a waiting list for any solid organ transplants.
13. Subject has previously received or scheduled to receive radiotherapy to coronary artery (brachytherapy), or chest/mediastinum.
14. Subject is receiving or will require chronic anticoagulation therapy (e.g., coumadin or any other agent for any reason).
15. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
16. Subject has a documented or suspected cirrhosis of Child-Pugh ≥ Class B.
17. Subject has known renal insufficiency;

    * Dialysis at the time of screening.
    * An estimated Glomerular filtration rate (GFR) < 30 ml/min/1.73m2
18. Subject is high risk of bleeding, or difficult to have appropriate treatment;

    * Has a history of bleeding diathesis or coagulopathy
    * Has had a significant gastro-intestinal or significant urinary bleed within the past six months
    * Has prior intracranial bleed
    * Has prior intracranial bleed (including severe permanent neurologic deficit that seem to be caused by previous intracranial bleeding)
    * Has known intracranial pathology that may cause intracranial bleeding per an investigator assessment (e.g. untreated aneurysm > 5 mm, arteriovenous malformation)
    * Subject will refuse blood transfusions
19. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months,
20. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
21. Subject has life expectancy < 3 year.
22. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
23. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
24. Subject whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g. subordinate hospital staff or sponsor staff) or subject is unable to read or write.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Kyoto University
Locations (39):
- Japan (39):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Fujita Health University, Toyoake-shi, Aichi-ken
  - ShinTokyo, Matsudo-shi, Chiba
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Kurume University, Kurume-shi, Fukuoka
  - Shinkoga Hospital, Kurume-shi, Fukuoka
  - Hanaoka Seishu Memorial Cardiovascular Clinic, Sapporo, Hokkaido
  - Kyoto University, Kyoto, Honshu
  - Kansairosai Hospital, Amagasaki-shi, Hyōgo
  - Kobe University, Kobe, Hyōgo
  - Tsukuba Medical Center, Tsukuba, Ibaraki
  - Iwate Medical University, Morioka, Iwate
  - Tokai University, Isehara-shi, Kanagawa
  - Shonankamakura General Hospital, Kamakura-shi, Kanagawa
  - Kanto Rosai Hospital, Kawasaki-shi, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Miyazak Medical Association Hospital, Miyazaki, Miyazaki
  - Tenri Hospital, Tenri-shi, Nara
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka University, Suita-shi, Osaka
  - The National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Saitama Medical Center Jichi Medical University, Saitama-shi, Saitama
  - Saitama Sekishinkai, Sayama-shi, Saitama
  - Juntendo University, Bunkyo-ku, Tokyo
  - University of Tokyo, Bunkyo-ku, Tokyo
  - Mitsui Memorial Museum, Chiyoda-ku, Tokyo
  - Sakakibara Memorial Hospital, Fuchu-shi, Tokyo
  - Teikyo University, Itabashi-Ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - The Cardiovascular Institute Hospital, Minato-Ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo
  - Dokkyo University, Tochigi, Utsunomiya
  - Wakayama Medical University Hospital, Kimiidera, Wakayama
  - Yamaguchi University, Ube-shi, Yamaguchi
  - Tokushima Red Cross Hospital, Tokushima
  - Abbott Vascular Japan Co., Ltd., Tokyo

REFERENCES:
- [Derived] Nishi T, Okada K, Kitahara H, Kameda R, Ikutomi M, Imura S, Hollak MB, Yock PG, Popma JJ, Kusano H, Cheong WF, Sudhir K, Fitzgerald PJ, Ellis SG, Kereiakes DJ, Stone GW, Honda Y, Kimura T; ABSORB III and ABSORB Japan Investigators. Intravascular ultrasound predictors of long-term outcomes following ABSORB bioresorbable scaffold implantation: A pooled analysis of the ABSORB III and ABSORB Japan trials. J Cardiol. 2021 Sep;78(3):224-229. doi: 10.1016/j.jjcc.2021.03.005. Epub 2021 Apr 21. PMID 33893022
- [Derived] Kozuma K, Tanabe K, Hamazaki Y, Okamura T, Ando J, Ikari Y, Nakagawa Y, Kusano H, Ediebah D, Kimura T; ABSORB Japan Investigators. Long-Term Outcomes of Absorb Bioresorbable Vascular Scaffold vs. Everolimus-Eluting Metallic Stent - A Randomized Comparison Through 5 Years in Japan. Circ J. 2020 Apr 24;84(5):733-741. doi: 10.1253/circj.CJ-19-1184. Epub 2020 Mar 26. PMID 32213737
- [Derived] Onuma Y, Honda Y, Asano T, Shiomi H, Kozuma K, Ozaki Y, Namiki A, Yasuda S, Ueno T, Ando K, Furuya J, Hanaoka KI, Tanabe K, Okada K, Kitahara H, Ono M, Kusano H, Rapoza R, Simonton C, Popma JJ, Stone GW, Fitzgerald PJ, Serruys PW, Kimura T. Randomized Comparison Between Everolimus-Eluting Bioresorbable Scaffold and Metallic Stent: Multimodality Imaging Through 3 Years. JACC Cardiovasc Interv. 2020 Jan 13;13(1):116-127. doi: 10.1016/j.jcin.2019.09.047. PMID 31918929
- [Derived] Stone GW, Kimura T, Gao R, Kereiakes DJ, Ellis SG, Onuma Y, Chevalier B, Simonton C, Dressler O, Crowley A, Ali ZA, Serruys PW. Time-Varying Outcomes With the Absorb Bioresorbable Vascular Scaffold During 5-Year Follow-up: A Systematic Meta-analysis and Individual Patient Data Pooled Study. JAMA Cardiol. 2019 Dec 1;4(12):1261-1269. doi: 10.1001/jamacardio.2019.4101. PMID 31561250
- [Derived] Okada K, Honda Y, Kitahara H, Otagiri K, Tanaka S, Hollak MB, Yock PG, Popma JJ, Kusano H, Cheong WF, Sudhir K, Fitzgerald PJ, Kimura T; ABSORB Japan Investigators. Bioresorbable Scaffold for Treatment of Coronary Artery Lesions: Intravascular Ultrasound Results From the ABSORB Japan Trial. JACC Cardiovasc Interv. 2018 Apr 9;11(7):648-661. doi: 10.1016/j.jcin.2017.11.034. PMID 29622143
- [Derived] Ali ZA, Gao R, Kimura T, Onuma Y, Kereiakes DJ, Ellis SG, Chevalier B, Vu MT, Zhang Z, Simonton CA, Serruys PW, Stone GW. Three-Year Outcomes With the Absorb Bioresorbable Scaffold: Individual-Patient-Data Meta-Analysis From the ABSORB Randomized Trials. Circulation. 2018 Jan 30;137(5):464-479. doi: 10.1161/CIRCULATIONAHA.117.031843. Epub 2017 Oct 31. PMID 29089314
- [Derived] Stone GW, Gao R, Kimura T, Kereiakes DJ, Ellis SG, Onuma Y, Cheong WF, Jones-McMeans J, Su X, Zhang Z, Serruys PW. 1-year outcomes with the Absorb bioresorbable scaffold in patients with coronary artery disease: a patient-level, pooled meta-analysis. Lancet. 2016 Mar 26;387(10025):1277-89. doi: 10.1016/S0140-6736(15)01039-9. Epub 2016 Jan 27. PMID 26825231
- [Derived] Kimura T, Kozuma K, Tanabe K, Nakamura S, Yamane M, Muramatsu T, Saito S, Yajima J, Hagiwara N, Mitsudo K, Popma JJ, Serruys PW, Onuma Y, Ying S, Cao S, Staehr P, Cheong WF, Kusano H, Stone GW; ABSORB Japan Investigators. A randomized trial evaluating everolimus-eluting Absorb bioresorbable scaffolds vs. everolimus-eluting metallic stents in patients with coronary artery disease: ABSORB Japan. Eur Heart J. 2015 Dec 14;36(47):3332-42. doi: 10.1093/eurheartj/ehv435. Epub 2015 Sep 1. PMID 26330419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target sample size was approximately 400 subjects (266 in the Absorb arm and 134 in the XIENCE arm) enrolled in approximately 40 investigational sites in Japan. First subject was enrolled on April 27, 2013 and the last subject completed 5-year follow-up on January 16, 2019.
Groups:
- Absorb BVS: Subjects receiving Absorb BVS
- XIENCE PRIME/XIENCE Xpedition: Subjects receiving XIENCE PRIME/XIENCE Xpedition
Period: Overall Study
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Started | 266 (Intent-to-treat (ITT) population) | 134 (Intent-to-treat (ITT) population)
Completed | 254 | 127
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition | Total
Number analyzed (Participants) | 266 | 134 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.4) | 67.3 (9.6) | 67.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 35 | 91
  Male | 210 | 99 | 309
Region of Enrollment [Number; unit: participants]
  Japan | 266 | 134 | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 1 year
Population: ITT population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 11 | 5

2. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

3. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

4. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 10 | 3

5. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 26 | 11

6. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 52 | 16

7. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 62 | 26

8. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 70 | 32

9. Secondary Outcome: Number of Participants With Any Death/Any MI/Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 74 | 34

10. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

11. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

12. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 9 | 3

13. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 16 | 7

14. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 29 | 9

15. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 34 | 11

16. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 40 | 14

17. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 10
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 41 | 17

18. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

19. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

20. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 8 | 3

21. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 19 | 5

22. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 23 | 7

23. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 27 | 9

24. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 28 | 10

25. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), un witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Myocardial Infarction (MI) Q wave MI: Development of new, pathological Q wave on the ECG. Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

26. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

27. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 8 | 3

28. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 9 | 3

29. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 15 | 4

30. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 17 | 4

31. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 18 | 7

32. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 25
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 20 | 8

33. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

34. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

35. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 1

36. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 13 | 6

37. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 25 | 10

38. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 31 | 12

39. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 37 | 14

40. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 33
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 38 | 17

41. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

42. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

43. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 1

44. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 13 | 5

45. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 24 | 7

46. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 28 | 9

47. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 34 | 10

48. Secondary Outcome: Number of Participants With Ischemia-driven TVR (ID-TVR)
Description: as for outcome 33
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 34 | 13

49. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the scaffold/stent.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

50. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

51. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 5 | 1

52. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 7 | 5

53. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 15 | 7

54. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 21 | 9

55. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 25 | 10

56. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 49
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 26 | 11

57. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: A revascularization is considered ischemia-driven if associated with any of the following:
  * Positive functional ischemia study including positive FFR
  * Ischemic symptoms and angiographic diameter stenosis ≥ 50% by core laboratory QCA
  * Angiographic diameter stenosis ≥ 70% by core laboratory QCA without angina or positive functional study
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

58. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

59. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 5 | 1

60. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 7 | 3

61. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 14 | 3

62. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 18 | 5

63. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 21 | 5

64. Secondary Outcome: Number of Participants With Ischemia-driven Revascularization (ID-TLR)
Description: as for outcome 57
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 21 | 6

65. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: Cardiac Death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all study procedure related deaths including those related to concomitant treatment.
  Vascular Death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular Death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

66. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 0 | 0

67. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 1 | 0

68. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 2 | 0

69. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 4 | 0

70. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 7 | 2

71. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 10 | 2

72. Secondary Outcome: Number of Participants Experiencing All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 65
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 15 | 4

73. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

74. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

75. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 8 | 3

76. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 9 | 3

77. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 14 | 4

78. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 16 | 4

79. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 17 | 7

80. Secondary Outcome: Number of Participants With All Myocardial Infarction ((MI: Q-wave Myocardial Infarction (Q-MI) or Non- Q-wave Myocardial Infarction (NQ-MI))
Description: as for outcome 73
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 19 | 7

81. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: ≤ 7 days post index procedure (In-hospital )
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 3 | 1

82. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 6 | 2

83. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 7 | 3

84. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants | 9 | 3

85. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 261 | 130
Participants | 13 | 4

86. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 258 | 128
Participants | 14 | 4

87. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 255 | 127
Participants | 15 | 6

88. Secondary Outcome: Number of Participants With Target Vessel MI (TV-MI)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 17 | 6

89. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: ITT population. Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  * Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation
  * Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation
  * Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation
  * Very late scaffold/stent thrombosis: >1 year post stent implantation
Time Frame: Acute (≤ 1 day)
Population: Stent/scaffold thrombosis event rates were determined according to the the analysis population with excluding subjects who are lost to follow-up through given time point without any Stent/Scaffold Thrombosis event.
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 266 | 133
Participants
  Definite | 0 | 0
  Probable | 0 | 0

90. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Subacute (>1 - 30 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 265 | 133
Participants
  Definite | 3 | 1
  Probable | 0 | 0

91. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Late (31 - 365 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 262 | 133
Participants
  Definite | 1 | 0
  Probable | 0 | 1

92. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Very Late (366 - 730 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 256 | 130
Participants
  Definite | 4 | 0
  Probable | 0 | 0

93. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Very Late (731 - 1095 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 249 | 126
Participants
  Definite | 1 | 0
  Probable | 0 | 0

94. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Very Late (1096 - 1460 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 240 | 125
Participants
  Definite | 0 | 0
  Probable | 0 | 0

95. Secondary Outcome: Number of Participants With Stent/Scaffold Thrombosis
Description: as for outcome 89
Time Frame: Very Late (1461 - 1825 days)
Population: as for outcome 89
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 234 | 122
Participants
  Definite | 0 | 0
  Probable | 0 | 0

96. Secondary Outcome: In-segment Late Loss (Non-inferiority)
Time Frame: 13 months
Population: Full Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 260 | 129
Participants | 5 | 5

97. Secondary Outcome: Nitrate Vaso-reactivity Analysis / In-device Mean Lumen Diameter : Pre-Nitroglycerin (NTG)
Description: Intracoronary nitrate injection was used for evaluating vaso-reactivity as it is routinely used during percutaneous coronary intervention (PCI) procedure.
Time Frame: 2 years
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: millimetre
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 82 | 43
millimetre | 2.43 (0.52) | 2.76 (0.52)

98. Secondary Outcome: Nitrate Vaso-reactivity Analysis/ In-device Mean Lumen Diameter: Absolute Vaso Dilatation
Description: Intracoronary nitrate injection was used for evaluating vaso-reactivity as it is routinely used during percutaneous coronary intervention (PCI) procedure.
  Absolute Vaso dilatation = Post Nitroglycerin (NTG) - Pre Nitroglycerin (NTG)
Time Frame: 2 years
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: millimetre
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 82 | 43
millimetre | 0.06 (0.14) | 0.07 (0.17)

99. Secondary Outcome: Nitrate Vaso-reactivity Analysis / In-device Mean Lumen Diameter : Post-Nitroglycerin (NTG)
Description: as for outcome 97
Time Frame: 2 years
Population: Full Analysis Set Population
Measure: Mean (Standard Deviation); unit: millimetre
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 82 | 43
millimetre | 2.49 (0.54) | 2.82 (0.54)

100. Secondary Outcome: Number of Participants With Cardiac Death, All MI, ID-TLR (MACE)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 30 | 11

101. Secondary Outcome: Number of Participants With Not Ischemia-driven TLR (NID-TLR)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 6 | 7

102. Secondary Outcome: Number of Participants With Non-Target Vessel MI (NTV-MI)
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
Number analyzed (Participants) | 254 | 127
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Absorb BVS | XIENCE PRIME/XIENCE Xpedition
All-Cause Mortality (participants affected / at risk) | 15/254 | 4/127
Serious Adverse Events (participants affected / at risk) | 127/266 | 61/134
Other Adverse Events (participants affected / at risk) | 217/266 | 110/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=266) | XIENCE PRIME/XIENCE Xpedition (N=134)
ANGINA PECTORIS (Cardiac disorders) | 9 | 4
ANGINA UNSTABLE (Cardiac disorders) | 1 | 3
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 2
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 9 | 3
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 16 | 11
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 0 | 1
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 12 | 3
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 5 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
POSTINFARCTION ANGINA (Cardiac disorders) | 1 | 0
PRINZMETAL ANGINA (Cardiac disorders) | 1 | 1
SINUS ARREST (Cardiac disorders) | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 | 1
VERTIGO (Ear and labyrinth disorders) | 2 | 1
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 | 2
CATARACT (Eye disorders) | 8 | 3
CORNEAL DEGENERATION (Eye disorders) | 1 | 0
DIABETIC RETINOPATHY (Eye disorders) | 2 | 0
EYELID PTOSIS (Eye disorders) | 1 | 0
MACULAR FIBROSIS (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 2 | 3
ENTERITIS (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 6 | 2
PERIODONTITIS (Gastrointestinal disorders) | 1 | 1
RECTAL POLYP (Gastrointestinal disorders) | 1 | 0
DISUSE SYNDROME (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1
PYREXIA (General disorders) | 1 | 1
THROMBOSIS IN DEVICE (General disorders) | 9 | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
DIABETIC GANGRENE (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 21 | 8
FALL (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 7 | 4
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 | 0
ELECTROCARDIOGRAM T WAVE PEAKED (Investigations) | 1 | 0
TRANSAMINASES INCREASED (Investigations) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 3
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL LIGAMENT OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
GASTRIC CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 7 | 3
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
HYPOGLYCAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
INTRACRANIAL HYPOTENSION (Nervous system disorders) | 0 | 1
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 3 | 1
THALAMUS HAEMORRHAGE (Nervous system disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 2 | 0
AORTIC RUPTURE (Vascular disorders) | 1 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 | 1
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 3 | 1
REPERFUSION INJURY (Vascular disorders) | 1 | 0
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb BVS (N=266) | XIENCE PRIME/XIENCE Xpedition (N=134)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 33 | 12
ANGINA UNSTABLE (Cardiac disorders) | 1 | 3
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 1 | 0
ARTERIOSPASM CORONARY (Cardiac disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 2
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 2
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 12 | 4
CORONARY ARTERY DISSECTION (Cardiac disorders) | 6 | 1
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 0 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 3 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 20 | 13
IN-STENT CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 0 | 1
INTRACARDIAC THROMBUS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 13 | 4
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 7 | 2
PALPITATIONS (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
POSTINFARCTION ANGINA (Cardiac disorders) | 1 | 0
PRINZMETAL ANGINA (Cardiac disorders) | 1 | 1
SINUS ARREST (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 | 2
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 3 | 2
VERTIGO (Ear and labyrinth disorders) | 4 | 1
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 1
PITUITARY HAEMORRHAGE (Endocrine disorders) | 0 | 1
STEROID WITHDRAWAL SYNDROME (Endocrine disorders) | 1 | 0
AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 1 | 0
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 0 | 2
CATARACT (Eye disorders) | 9 | 3
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 1 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 1 | 1
CORNEAL DEGENERATION (Eye disorders) | 1 | 0
DIABETIC RETINOPATHY (Eye disorders) | 2 | 0
EYELID PTOSIS (Eye disorders) | 2 | 0
MACULAR FIBROSIS (Eye disorders) | 1 | 0
MACULAR OEDEMA (Eye disorders) | 1 | 0
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 1 | 0
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0
ABDOMINAL WALL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
CHEILITIS (Gastrointestinal disorders) | 1 | 0
COLONIC POLYP (Gastrointestinal disorders) | 6 | 4
CONSTIPATION (Gastrointestinal disorders) | 7 | 2
DENTAL CARIES (Gastrointestinal disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 0
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 2 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 5 | 0
GASTRITIS ATROPHIC (Gastrointestinal disorders) | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 3 | 1
ILEUS (Gastrointestinal disorders) | 1 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 6 | 2
MELAENA (Gastrointestinal disorders) | 1 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0
PAROTID GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 | 1
PERIODONTITIS (Gastrointestinal disorders) | 2 | 1
RECTAL POLYP (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1
ADVERSE DRUG REACTION (General disorders) | 10 | 3
CATHETER SITE HAEMATOMA (General disorders) | 3 | 2
CATHETER SITE HAEMORRHAGE (General disorders) | 2 | 1
CATHETER SITE PAIN (General disorders) | 2 | 2
CATHETER SITE RASH (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 10 | 10
DISUSE SYNDROME (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0
INJECTION SITE PHLEBITIS (General disorders) | 1 | 0
MALAISE (General disorders) | 3 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 6 | 4
OEDEMA PERIPHERAL (General disorders) | 6 | 0
PYREXIA (General disorders) | 1 | 1
THROMBOSIS IN DEVICE (General disorders) | 9 | 1
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 2 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
ANAPHYLACTOID REACTION (Immune system disorders) | 1 | 0
CONTRAST MEDIA ALLERGY (Immune system disorders) | 3 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 1
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 2 | 0
CYSTITIS (Infections and infestations) | 0 | 2
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
DIABETIC GANGRENE (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 4 | 0
HERPES ZOSTER (Infections and infestations) | 4 | 0
HORDEOLUM (Infections and infestations) | 2 | 0
INFLUENZA (Infections and infestations) | 4 | 1
NASOPHARYNGITIS (Infections and infestations) | 27 | 14
PHARYNGITIS (Infections and infestations) | 1 | 1
PNEUMONIA (Infections and infestations) | 3 | 0
PYODERMA (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 1
TINEA INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 1
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 2
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 7 | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 21 | 8
FALL (Injury, poisoning and procedural complications) | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 7 | 4
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0
OPEN WOUND (Injury, poisoning and procedural complications) | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 40 | 17
BLOOD CREATINE PHOSPHOKINASE MB INCREASED (Investigations) | 19 | 12
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 | 0
BLOOD PRESSURE DECREASED (Investigations) | 3 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 1
CARDIAC ENZYMES INCREASED (Investigations) | 13 | 5
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 1
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 5 | 1
ELECTROCARDIOGRAM T WAVE PEAKED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 3 | 1
N-TERMINAL PROHORMONE BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 1 | 0
OCCULT BLOOD POSITIVE (Investigations) | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 1 | 0
TROPONIN I INCREASED (Investigations) | 3 | 3
WEIGHT DECREASED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 8 | 10
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 3 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 3
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
SERONEGATIVE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 3 | 0
SPINAL LIGAMENT OSSIFICATION (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ANGIOIMMUNOBLASTIC T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
GASTRIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
GASTRIC CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 7 | 3
CERVICAL MYELOPATHY (Nervous system disorders) | 1 | 0
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 | 0
CHOLINERGIC SYNDROME (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 2 | 1
DIZZINESS POSTURAL (Nervous system disorders) | 0 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 3 | 2
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
HYPOGLYCAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 | 0
INTRACRANIAL HYPOTENSION (Nervous system disorders) | 0 | 1
NEURALGIA (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 2
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 0
SCIATICA (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 3 | 2
TENSION HEADACHE (Nervous system disorders) | 1 | 0
THALAMUS HAEMORRHAGE (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
HEAD BANGING (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 4 | 3
NEUROSIS (Psychiatric disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 2 | 1
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 1 | 0
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 3 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1
POLLAKIURIA (Renal and urinary disorders) | 2 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 1
URATE NEPHROPATHY (Renal and urinary disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 1
HAEMATOSPERMIA (Reproductive system and breast disorders) | 1 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 0
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 2
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ALKALOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY TRACT HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 | 0
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 5 | 0
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC BULLOSIS (Skin and subcutaneous tissue disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 2 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 5 | 2
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 0 | 1
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 3
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 | 2
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
PARAPSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURIGO (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 4 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0
SENILE PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
TOOTH EXTRACTION (Surgical and medical procedures) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 2 | 0
AORTIC RUPTURE (Vascular disorders) | 1 | 0
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
EXTRAVASATION BLOOD (Vascular disorders) | 0 | 1
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 7 | 5
HYPOTENSION (Vascular disorders) | 1 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 3 | 1
PERIPHERAL COLDNESS (Vascular disorders) | 2 | 0
REPERFUSION INJURY (Vascular disorders) | 1 | 1
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 | 0
VARICOPHLEBITIS (Vascular disorders) | 1 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes